# **Clinical Development**

Clinical Trial Protocol ID: IRB\_00138483

# IMPROVING HEALTH INSURANCE LITERACY AMONG UTAH'S HISPANIC COMMUNITY

Principal or Coordinating Investigator: Anne Kirchhoff

| Site Name | Investigator | Staff Name(s) |
|---|---|---|
| University of Utah/Huntsman Cancer<br>Institute | Anne Kirchhoff | Heydon Kaddas |
| | | Austin Waters |
| | | Perla Vaca Lopez |
| | | Judy Ou |
| | | Karely van Thiel Berghuijs |
| Site Name | Investigator | Staff Name(s) |
| Utah Health Policy Project | Anne Kirchhoff | Heydon Kaddas |
| | | Austin Waters |
| | | Perla Vaca Lopez |
| | | Judy Ou |
| | | Karely van Thiel Berghuijs |

Document type: Draft Protocol Summary

Version number: v3

Release date: 10.4.23

# **Table of Contents**

| Clinical Development | |
|----------------------------------------------------------|----------|
| Protocol Synopsis | 3 |
| Amendments | <i>6</i> |
| 1. Background and Introduction | 7 |
| 2. Purpose and Objectives | ε |
| 3. Study Population | g |
| 3.1 Inclusion Criteria: | 9 |
| 3.2 Exclusion Criteria: | 9 |
| 4. Study design | 10 |
| 5. Study Procedures | 10 |
| 5.1 Recruitment/Participant Identification Process | 10 |
| 5.2 Informed Consent | 11 |
| 5.3 Study duration | 11 |
| 5.4 Randomization | 11 |
| 5.5 Procedures | 11 |
| 6. Data Collection | 11 |
| 7. Risks and Benefits | 12 |
| 8. Cost and Compensation | 13 |
| 9. Statistical Methods, Data Analysis and Interpretation | 13 |
| 9.1 Aim 2 | 14 |
| 9.2 Aim 3 | 15 |
| Poforoncos | 1/ |

# **Protocol Synopsis**

| Protocol number | 00138483 |
|---|---|
| Title | IMPROVING HEALTH INSURANCE LITERACY AMONG UTAH'S HISPANIC COMMUNITY |
| Sponsor and Clinical Phase | The National Center for Advancing Translational Sciences of the National Institutes of Health, Award Number(s) UL1TR002538 |
| Study type | |
| Primary Objective(s) | We woonducted with the purpose of gaining feedback on an existing health insurance education program (HIEP), originally created for young adult cancer patients. We will do this by the following study aims: Aim 2. Pilot test the HIEP with Hispanic community members to further refine the intervention and evaluate its efficacy. |
| Study design | Non-Experimental and/or Descriptive Research Design • Survey/Questionaire Research Experimental and/or Interventional Research Design • Prospective social/ Behavioral Intervention or Experiment |
| Population | Hispanic community members |
| Inclusion criteria | -18-64 years of age -Self-identify as Hispanic -Speak English and or Spanish -Resident of Utah -Primary policyholder -Recently enrolled in any kind of health insurance within the past year |
| Exclusion criteria | <ul> <li>Younger than 18 years of age</li> <li>Hispanic Community Members:</li> <li>Not Hispanic of Latinx in origin</li> <li>Key Informants:</li> <li>Work for an organization that does not serve the</li> <li>Hispanic or Latinx community</li> </ul> |

University of Utah
Protocol Version 03
Protocol No. 00138483

Data analysis

Analysis of the pre-post health literacy survey results: McNemar's tests will identify significant changes in the percent of questions answered correctly. We will utilize logistic regression models with generalized estimating equations to calculate the odds of improvement in health insurance literacy while accounting for within-person clustering. Models will control for acculturation and/or preferred language, current insurance status, sex, and age. We will stratify models to obtain group-specific effect estimates by current insurance status, sex, 10-year age groups, and employment status.


### **Amendment 4**

The amendment was necessary to remove personnel off the IRB who were no longer part of the team. The following sections reflected this change:

- 1. Contact and title Study introduction
- 2. Study Location and Sponsors
- 3. Study information consent process
- 4. Resources and Responsibilities

## **Amendment 3**

We submitted the translated (Spanish) version of approved documents: this includes submitting the consent, baseline, follow up survey, and outline of the education pilot program. We also added new study personnel. The following sections reflect this change

- 1. Documents and attachments
- 2. Section 2: Study Location & Sponsors

#### **Amendment 2**

Amendment 2 was necessary because we needed to add new study personnel. We also needed to change the inclusion criteria to be more specific to our target population for aim 2 and to increase recruitment efforts, we also included social media as a form of recruitment. The consent form also needed to be submitted for this aim. For quality purposed, we decided to also include for the pilot sessions to be recorded. Participate compensation for aim 2 was decreased. Funding for the project ended and we needed to remove the sponsor from the study. We also increased the timeframe of the study since more time is needed to complete the study. The following sections reflect this change:

- 1. Study location and sponsors (Section 1, section 3)
- 2. Participants (section 5)
- 3. Study information (section 3, section 4a, section 4b, and section 6)
- 4. Consent process (Section 1)
- 5. Risk and Benefits (Section 4a and section 4c)
- 6. Data Monitoring Plan (Section 5)
- 7. Resources & Responsibilities (Section 1)
- 8. Documents and Attachments

### **Amendment 1**

Translation of approved study documents needed to be submitted since a substantial portion of participants will be Spanish speaking.

University of Utah Protocol Version 03

1. Study information - Consent Process, Documents and attachments.


## 1. Background and Introduction

The 2010 Patient Protection and Affordable Care Act (ACA) increased health insurance coverage nationally by providing subsidies to lower insurance costs and expanding Medicaid. Through the ACA, funding was earmarked for health insurance navigators at community organizations to assist uninsured individuals in enrolling for coverage through the Health Insurance Marketplaces and Medicaid. In Utah, the **Utah Health Policy Project (UHPP)** is a trusted community resource, focused on advancing sustainable health care solutions for underserved Utahns through better access, education, and public policy. UHPP frequently works with the Hispanic community, who comprise 80% of the clients they serve. UHPP enrollment efforts have been stymied in recent years due to federal budget cuts that defunded health insurance navigators and the lack of state resources available to replenish cuts to the health insurance navigator program.

The goal of our CCTS project is to create materials to improve health insurance literacy for UHPP's Hispanic clients. Health insurance literacy is one's ability to make informed decisions about choosing and using health insurance. By providing Hispanic community members with resources to improve their understanding of insurance, this effort can help to address the gaps in navigation services and allow them to make informed decisions about selecting and using their insurance coverage. In this grant, we will adapt materials for Hispanic community members from Dr. Kirchhoff's existing health insurance literacy program that was designed for cancer patients (NCI R01 (1R01CA242729). The content of the current literacy program includes information on insurance types (e.g., public vs. private), information on insurance cost sharing mechanisms (e.g., deductibles), an overview of health insurance laws including the ACA, and cost reduction strategies (e.g., understanding in- vs. out-of-network providers). However, the current program was not designed for a general population audience nor considering the cultural or linguistic needs of the Hispanic community. Thus, during the CCTS grant, we will adapt and pilot test the revised program with Hispanic community members recruited by the UHPP.


## 2. Purpose and Objectives

The purpose of this study is to adapt a health insurance education program to the Hispanic/Latinx population Utah's population.

Aim 2. Pilot test the HIEP with Hispanic community members to further refine the intervention and evaluate its efficacy. We will then refine the intervention by pilot testing the adapted intervention with Hispanic community members (n=10-15) recruited by UHPP. Pilot testing of the HIEP will be conducted to identify acceptability of content and potential implementation issue areas, as well as any discordance in cultural values, beliefs, or feelings about health insurance.

University of Utah Protocol Version 03

## 3. Study Population

Age of Participants: 18-64 years old

Sample Size: All Centers: 75

#### 3.1 Inclusion Criteria:

- -18-64 years of age
- -Self-identify as Hispanic
- -Speak English and or Spanish
- -Resident of Utah
- -Primary policyholder
- -Recently enrolled in any kind of health insurance within the past year

#### 3.2 Exclusion Criteria:

- Younger than 18 years of age

**Hispanic Community Members:** 

- Not Hispanic of Latinx in origin


## 4. Study design

Non-Experimental and/or Descriptive Research Design:

Survey/Questionnaire Research

Experimental and/or Interventional Research Design:

• Prospective social/behavioral intervention or experiment

## 5. Study Procedures

### **5.1 Recruitment/Participant Identification Process**

#### 5.1.1 Enrollment Goals

# Aim 2. Pilot test the HIEP with Hispanic community members to further refine the intervention and evaluate its efficacy.

Hispanic community members (n=10-15)

#### 5.1.2. Process

Prior to the beginning of recruitment for the interviews with Hispanic community members, the Kirchhoff Team and UHPP staff will work together to develop a culturally tailored survey in English and Spanish (which will be submitted for approval via an amendment). All documents will be translated from English to Spanish and submitted for IRB approval prior to recruitment of any participants. Participants will be identified through the recruitment methods outlined above.

#### Aim 2

- Once the intervention is adapted we will again work with UHPP to recruit additional new Hispanic community members to pilot test the intervention. Pilot testing will be conducted primarily by UHPP staff. Prior to the start of the pilot test, participants will be asked to consent using a consent cover letter. The pilot session will be recorded through Zoom or audio recorded with team recorders for fidelity purposes. Pilot testing will include a short pre-post survey to assess change in health insurance literacy. The post survey may also include a short audio recorded interview about the intervention and areas of improvement. Pilot activities will primarily be conducted by UHPP staff but may be conducted a member of the Kirchhoff team.
- Further refinement of the intervention materials and statistical analyses will be conducted by the Kirchhoff Team, again contextualized by UHPP.
- Feedback on the results of each phase of the study will be elicited from UHPP staff. The Kirchhoff team will then lead manuscript writing for each aspect of the study with assistance from UHPP. All members of the UHPP team mentioned above have been trained in Human Subjects


Research jointly by CCTS and the IRB and are present on this application.

#### 5.2 Informed Consent

Location(s) where consent will be obtained: Utah Health Policy Project Out in the community Over the phone Online

Description of the consent process(es), including the timing of consent: Study staff/UHPP staff/CCTS staff will reach out to referred participants to gauge interest in the study an obtain consent. There is no minimum amount of time between digital approach and consent as this study is quite minimal risk. Potential participants will be given as much or as little time to decide if they would like to participate as they would like. Study staff will be available throughout to answer any questions. The voluntary nature of research studies will be stressed when potential participants are approached. Participants will be informed prior to the start of the interview/engagement studio/pilot test that they may stop at any time and have the right not to answer any question. Potential participants will be allowed to schedule their interview/pilot test whenever they find appropriate and will be encouraged to ask questions to the study coordinator, before the interview/pilot testing is conducted.

## 5.3 Study duration

Study duration will be approximately 3 years

#### 5.5 Procedures

- Prior to the beginning of recruitment for the interviews with Hispanic community members, the Kirchhoff Team and UHPP staff will work together to develop a culturally tailored survey and interview script in English and Spanish (which will be submitted for approval via an amendment). All documents will be translated from English to Spanish and submitted for IRB approval prior to recruitment of any participants.
- Participants will be identified through the recruitment methods outlined above. Qualitative interviews and studio sessions will be conducted with the purpose of gaining feedback on an existing health insurance education program (HIEP), originally created for young adult cancer patients in the HIAYA CHAT Study.


- Once the intervention is adapted we will again work with UHPP to recruit additional new Hispanic community members to pilot test the intervention. Pilot testing will be conducted primarily by UHPP staff. Prior to the start of the pilot test, participants will be asked to consent using a consent cover letter. The pilot session will be recorded through Zoom or audio recorded with team recorders for fidelity purposes. Pilot testing will include a short pre-post survey to assess change in health insurance literacy. The post survey may also include a short audio recorded interview about the intervention and areas of improvement. Pilot activities will primarily be conducted by UHPP staff but may be conducted a member of the Kirchhoff team.
- Further refinement of the intervention materials and statistical analyses will be conducted by the Kirchhoff Team, again contextualized by UHPP.
- Feedback on the results of each phase of the study will be elicited from UHPP staff. The Kirchhoff team will then lead manuscript writing for each aspect of the study with assistance from UHPP. All members of the UHPP team mentioned above have been trained in Human Subjects Research jointly by CCTS and the IRB and are present on this application.

#### 6. Data Collection

The team will use the Research Electronic Data Capture (REDCap) software application to collect and manage the data for this project. The REDCap database is on a secure server maintained by the Huntsman Cancer Institute (HCI) bioinformatics shared resource and the HCI Computer and Technology Group (CATG).

Voice recordings will be stored securely on the Kirchhoff Team drive at Huntsman Cancer Institute or on password protected computers at HCI.

## 7. Risks and Benefits

- The potential risks to participants are minimal. Participants may feel slight psychological distress when answering questions about health insurance and cost concerns.
- There is also a risk of breach of confidentiality of the participants.
- No direct benefit. From the societal perspective though, the benefits include improved knowledge about the Hispanic perceptions of health insurance.

rotocol Version 03 Protocol No. 00138483

## 8. Cost and Compensation

- There is no cost to be in this study
- There will be gift card compensation available for participants,
  - Pilot testing pre and post surveys: \$40

## 9. Statistical Methods, Data Analysis and Interpretation

Further refinement of the intervention materials and statistical analyses will be conducted by the Kirchhoff Team, again contextualized by UHPP.

Feedback on the results of each phase of the study will be elicited from UHPP staff. The Kirchhoff team will then lead manuscript writing for each aspect of the study with assistance from UHPP. All members of the UHPP team mentioned above have been trained in Human Subjects Research jointly by CCTS and the IRB and are present on this application.

Analysis of the pre-post health literacy survey results: McNemar's tests will identify significant changes in the percent of questions answered correctly before and after intervention. We examine differences in Health Insurance Literacy Measure before and after intervention. We will stratify this variable by age and language spoken.

## References

- 1. Noe-Bustamante L, Lopez MH, Krogstad JM. *U.S. Hispanic population surpassed 60 million in 2019, but growth has slowed.* Pew Research Center;2020.
- 2. Kem C. Gardner Policy Institute. *U.S. Census Bureau Estimates for Race and Hispanic Origin, Vintage 2019.* University of Utah David Eccles School of Business Kem C. Gardner Policy Institute;2020.
- 3. Aragones A, Hayes SL, Chen MH, González J, Gany FM. Characterization of the Hispanic or latino population in health research: a systematic review. *Journal of immigrant and minority health*. 2014;16(3):429-439.
- 4. Foundation KF. Uninsured Rates for the Nonelderly by Race/Ethnicity. 2019; https://www.kff.org/uninsured/state-indicator/nonelderly-uninsured-rate-by-raceethnicity/?currentTimeframe=0&sortModel=%7B%22colId%22:%22Black%22,%22sort%22:%22desc%22%7D. Accessed 11/11/2020.
- 5. Obama B. United States Health Care Reform: Progress to Date and Next Steps. *JAMA*: the journal of the American Medical Association. 2016;316(5):525-532.
- 6. French MT, Homer J, Gumus G, Hickling L. Key Provisions of the Patient Protection and Affordable Care Act (ACA): A Systematic Review and Presentation of Early Research Findings. *Health services research.* 2016;51(5):1735-1771.
- 7. Courtemanche C, Marton J, Ukert B, Yelowitz A, Zapata D. Early Impacts of the Affordable Care Act on Health Insurance Coverage in Medicaid Expansion and Non-Expansion States. *Journal of Policy Analysis and Management.* 2017;36(1):178-210.
- 8. Clemans-Cope L, Long SK, Coughlin TA, Yemane A, Resnick D. The Expansion of Medicaid Coverage under the ACA: Implications for Health Care Access, Use, and Spending for Vulnerable Low-income Adults. *Inquiry*. 2013;50(2):135-149.
- 9. Buchmueller TC, Levy HG. The ACA's Impact On Racial And Ethnic Disparities In Health Insurance Coverage And Access To Care. *Health Affairs*. 2020;39(3):395-402.
- 10. Pollitz K, Tolbert J. *Data Note: Limited Navigator Funding for Federal Marketplace States.* Kaiser Family Foundation;2020.
- 11. Pérez-Escamilla R, Garcia J, Song D. HEALTH CARE ACCESS AMONG HISPANIC IMMIGRANTS: ¿ALGUIEN ESTÁ ESCUCHANDO? [IS ANYBODY LISTENING?]. NAPA Bull. 2010;34(1):47-67.
- 12. States NRCUPoHitU. Access to and Quality of Health Care. In: Tienda M, Mitchell F, eds. *Hispanics and the Future of America*. Vol 10. Washington DC: National Academies of Press; 2006.
- 13. Ghaddar S, Byun J, Krishnaswami J. Health insurance literacy and awareness of the Affordable Care Act in a vulnerable Hispanic population. *Patient Education and Counseling*. 2018;101(12):2233-2240.
- 14. Krogstad JM, Gonzalez-Barrera A, Noe-Bustamante L. *U.S. Latinos among hardest hit by pay cuts, job losses due to coronavirus*. Online: Pew Research Center;2020.
- 15. Hofstede G. *Culture's consequences: Comparing values, behaviors, institutions and organizations across nations.* Vol 2nd. Thousand Oaks, CA: Sage; 2001.
- 16. Hall ET. *Beyond culture*. Garden City, NY: Anchor Press; 1976.
- 17. Paez KA, Mallery CJ, Noel H, et al. Development of the Health Insurance Literacy Measure (HILM): conceptualizing and measuring consumer ability to choose and use private health insurance. *Journal of health communication*. 2014;19 Suppl 2:225-239.
- 18. Marin G, Sabogal F, Marin BV, Otero-Sabogal R, Perez-Stable EJ. Development of a Short Acculturation Scale for Hispanics. *Hispanic Journal of Behavioral Sciences*. 1987;9(2):183-205.
- 19. Wu YP, Thompson D, Aroian KJ, McQuaid EL, Deatrick JA. Commentary: Writing and Evaluating Qualitative Research Reports. *Journal of pediatric psychology*. 2016;41(5):493-505.


- 20. Elo S, Kyngas H. The qualitative content analysis process. *Journal of advanced nursing*. 2008;62(1):107-115.
- 21. Saldana J. The Coding Manual for Qualitative Researchers. London, UK: Sage Publishing; 2013.